CLINICAL TRIAL: NCT01316029
Title: A Large Cross-sectional Study of Laying-on-of-hands in Japan: Who Responds to it and What Facilitates the Response?
Brief Title: Safety/Effectiveness Study of a Single Session of Laying-on-of-hands in Various Settings in Japan
Acronym: SELH
Status: Completed | Type: Observational
Sponsor: MOA Health Science Foundation (Other)
Responsible Party: Yukio Yagisawa, MOA Health Science Foundaiton
Other Study IDs: MHS-001
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2007-01

CONDITIONS: Signs and Symptoms; Physical Disorders; Personal Satisfaction
Keywords: Laying-on-of-hands; Therapeutic touch; cross-sectional study; healing environment; safety and effectiveness; optimal condition for the intervention
MeSH Terms: conditions — Signs and Symptoms; Personal Satisfaction | interventions — Therapeutic Touch

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- laying-on-of-hands: 44,587 Japanese volunteers with/without illness, who were interested in receiving laying-on-of-hands
  Interventions: Procedure: Okada Purifying Therapy

INTERVENTIONS:
Procedure: Okada Purifying Therapy — Each participant received a single session of Okada Purifying Therapy lasting 30 minutes or longer, administered by a voluntary certified practitioner.
  Other Names: laying-on-of-hands; biofield therapy; Therapeutic touch

SUMMARY:
The purpose of this study is to determine the symptomatic changes after a single session of laying-on-of-hands in various settings, and to evaluate optimal conditions for the outcomes.

DETAILED DESCRIPTION:
Laying-on-of-hands is applied in many different situations; however, most reports published previously described its efficacy in a clinical setting, with its administration conducted by a few expert practitioners. This study aimed to determine the symptomatic changes after a single session of the Okada Purifying Therapy, a form of laying-on-of-hands, in various settings, and to analyze factors influencing the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* able to receive laying-on-of-hands for 30 minutes or longer from the investigators
* able to self-evaluate the change of their symptoms
* competent to answer the Japanese questionnaires
* aged 16 years or older

Exclusion Criteria:

* those who did not match the inclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any Japanese people who were interested in receiving laying-on-of-hands
Sampling Method: Non-Probability Sample
Enrollment: 44587 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Severity of various symptoms | Baseline and immediately after a single intervention
  Participants self-evaluated the severity of various symptoms before and after the intervention, and determined whether their symptoms got better, worsened, or did not change.

SECONDARY OUTCOMES:
Adjusted odds ratios of the factors influencing the outcomes | in 1 year
  After collecting all the eligible data, to be clarified are such personal variables as demographic attributes associated with the tendency to respond, and factors that facilitate such responses.

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoshi Suzuki, MD, PhD, Principal Investigator — MOA Health Science Foundation
Locations (1):
- MOA Health Science Foundation, Tokyo, Tokyo, Japan

REFERENCES:
- See also: Click here for more information about activities of MOA Health Science Foundation (Japanese) — http://www.mhs.or.jp
- See also: Click here for more information about Okada Purifying Therapy, a laying-on-of-hands. — http://www.moainternational.or.jp